CLINICAL TRIAL: NCT06246305
Title: The Effect of Virtual Reality Intervention and Its Impact on Upper Extremity Function in Patients With Post-operative Rotator Cuff Repair
Brief Title: Effect of Virtual Reality on Upper Extremity Function Post-operative Rotator Cuff Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed ElMelhat, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VR on rotator cuff repair
Record Dates: First submitted 2024-01-27; First posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-01

CONDITIONS: Rotator Cuff Impingement Syndrome; Rotator Cuff Tears; Rotator Cuff Injuries
Keywords: rotator cuff repair; post-operative; upper extremity; function
MeSH Terms: conditions — Shoulder Impingement Syndrome; Rotator Cuff Injuries

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into one of the 2 groups: the control group receiving the conventional physical therapy intervention or to the experimental group receiving virtual reality intervention
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional physical therapy (Active Comparator): The conventional therapy rehabilitation program is divided into three phases: on-brace, off-brace, and active mobilization. The on-brace phase (post-op 0-6 weeks) mainly consists of low-intensity whole-body exercises with shoulder girdle, elbow, and hand mobilization exercises on the affected side. In this phase, exercises are done of three sets with 10 repetitions per day. The off-brace phase (post-op 6-9 weeks) consists of passive shoulder ROM exercises using an exercise stick and an early scapular stabilization exercise. The active mobilization phase (post-op 9-12 weeks) consists of both active and passive shoulder ROM , strengthening exercise with progressive resistance using TheraBand, and scapular stabilization exercises. During the off-brace and active mobilization phases, exercises are done of 3-5 sets of exercises with 10 repetitions per day.
  Interventions: Other: conventional physical therapy training
- Virtual reality (VR) (Experimental): During the on-brace phase(0-6 weeks), participants in this group will use the program as performed in the control group. During the off-brace (6-9 weeks post-op) and active mobilization phases (9-12 weeks post-op), participants will use the Virtual Reality machine. This program includes warming and cooling periods with posterior, anterior and inferior capsule stretching and pectoral muscle stretching. Exercise training includes bilateral shoulder elevation, boxing, bowling and tennis games accompanied by avatar. Resistance training is progressed in the active mobilization phase using TheraBand.
  Interventions: Device: Virtual Reality (VR) training

INTERVENTIONS:
Other: conventional physical therapy training — conventional therapy rehabilitation program is divided into three phases: on-brace, off-brace, and active mobilization. The on-brace phase (post-op 0-6 weeks) mainly consists of low-intensity whole-body exercises with shoulder girdle, elbow, and hand mobilization exercises on the affected side. The off-brace phase (post-op 6-9 weeks) consists of passive shoulder ROM exercises using an exercise stick and an early scapular stabilization exercise. The active mobilization phase (post-op 9-12 weeks) consists of both active and passive shoulder ROM , strengthening exercise with progressive resistance, and scapular stabilization exercises. The intervention is done 3 times per week for 12 weeks.
  Arms: Conventional physical therapy
Device: Virtual Reality (VR) training — During the on-brace phase (0-6 weeks), participants in this group will use the program as performed in the control group. During the off-brace (6-9 weeks post-op) and active mobilization phases (9-12 weeks post-op), participants will use the Virtual Reality machine. this program involves warming up and down stretching exercises and exercise training that includes bilateral shoulder elevation, boxing, bowling and tennis games accompanied by avatar. The intervention is done 3 times per week for 12 weeks.
  Arms: Virtual reality (VR)

SUMMARY:
The aim of the study is to investigate the effect and the impact of performing virtual reality intervention on upper extremity function in patients with post-operative rotator cuff repair. The main question that it aims to answer is:

Does the application of virtual reality intervention improves upper extremity function in patients with post-operative rotator cuff repair.

Participants will be randomized into 2 groups: the control group receiving conventional physical therapy intervention and the experimental group receiving the virtual reality intervention.

DETAILED DESCRIPTION:
Rotator cuff tears are one of the most common disorders of the shoulder that result in shoulder pain and dysfunction. It affects about 30% of individuals that are older than 60 years. The conservative management is the first-line treatment for a rotator cuff tear, but a surgical rotator cuff repair (RCR) is required if the conservative management failed. Post-operative rehabilitation requires up to 12 weeks. But, Virtual Reality (VR) intervention is emerging as a viable alternative for musculoskeletal rehabilitation of the upper limb. Unlike in neuro-rehabilitation, VR is still poorly used in orthopedic rehabilitation. Thus, the investigators hypothesize that performing virtual reality intervention will improve the upper extremity function in patients with post-operative rotator cuff repair.

ELIGIBILITY:
Inclusion Criteria:

1. Older than 18 years old and younger than 70 years old, and referred by the Adult Orthopedic Department with arthroscopic RC repair of a non-retracted isolated full-thickness supraspinatus tear with maximum 5 days post operation.
2. Poor response to initial non-operative treatment.

Exclusion Criteria:

1. Large-sized RC tears (3-5 cm),
2. Massive or irreparable RC tears,
3. Anteroinferior labral (Bankart) or superior labrum anterior to posterior lesions,
4. Severe glenohumeral osteoarthritis,
5. Adhesive capsulitis, or
6. Previous surgery on the affected shoulder
7. Re-tears of the RC.
8. Indication for revision RCR
9. Severe neurological deficits
10. Infection in the affected shoulder
11. Blindness and/or illiteracy

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-28 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Shoulder function with disabilities of arm, shoulder and hand | Measured at baseline, after 6 weeks, and after 12 weeks
  in numbers, it ranges from 0 to 100 with 0 being the lowest and 100 the highest. The higher the score means the better outcome

SECONDARY OUTCOMES:
The Numerical Pain Intensity Rating Scale | Measured at baseline, after 6 weeks, and after 12 weeks
  in numbers, it ranges from 0 to 10 with 0 being the lowest and 10 being the highest. The higher the score means the better outcome
Active and passive range of motion using goniometer | Measured at baseline, after 6 weeks, and after 12 weeks
  in degrees
Isometric muscle test by Handheld Dynamometer | Measured at baseline, after 6 weeks, and after 12 weeks
  in numbers, it ranges from 0 to 5 with 0 being the lowest and 5 the highest. The higher the score means the better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed El Melhat, PhD, Study Director — Cairo University
Locations (1):
- Ahmed ElMelhat [aelmelhat], Cairo, Egypt

REFERENCES:
- [Background] Gutierrez-Espinoza H, Araya-Quintanilla F, Pinto-Concha S, Zavala-Gonzalez J, Gana-Hervias G, Cavero-Redondo I, Alvarez-Bueno C. Effectiveness of supervised early exercise program in patients with arthroscopic rotator cuff repair: Study protocol clinical trial. Medicine (Baltimore). 2020 Jan;99(4):e18846. doi: 10.1097/MD.0000000000018846. PMID 31977882
- [Background] Correia FD, Molinos M, Luis S, Carvalho D, Carvalho C, Costa P, Seabra R, Francisco G, Bento V, Lains J. Digitally Assisted Versus Conventional Home-Based Rehabilitation After Arthroscopic Rotator Cuff Repair: A Randomized Controlled Trial. Am J Phys Med Rehabil. 2022 Mar 1;101(3):237-249. doi: 10.1097/PHM.0000000000001780. PMID 33935152
- See also: Post-operative rehabilitation using a digital healthcare system in patients who had undergone rotator cuff repair: protocol for a single-center randomized controlled trial — http://doi.org/10.1186/s13063-022-06648-4
- See also: A randomized controlled trial of postoperative rehabilitation using digital healthcare system after rotator cuff repair — http://doi.org/10.1038/s41746-023-00842-7
- See also: Comparison of virtual reality exergaming and home exercise programs in patients with subacromial impingement syndrome and scapular dyskinesis: Short term effect — http://doi.org/10.1016/j.aott.2017.03.008
- See also: The Effects of Virtual Reality Exergaming on Pain, Functionality and Acromiohumeral Distance in Shoulder Impingement Syndrome Patients: A Randomized Controlled Study — http://dx.doi.org/10.5336/healthsci.2020-74413